CLINICAL TRIAL: NCT05623748
Title: Establishment and Application of 3-Dimensional (3-D) Cell Culture Model of Clinical Circulating Tumor Cells (CTCs)
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101222A3
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cell Carcinoma
Keywords: CTCs; 3-D Cell culture; Cell purification; Cell proliferation
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer for CTC culture: participants are cancer patients with transitional cell carcinoma
  Interventions: Procedure: CTCs isolation/purification and cell number expansion
- Healthy for CTC culture: enroll participants without cancer
  Interventions: Procedure: CTCs isolation/purification and cell number expansion

INTERVENTIONS:
Procedure: CTCs isolation/purification and cell number expansion — In the 1st year research project, investigators will further validate and evaluate the clinical feasibility of using a 3-D cell culture model for CTCs isolation/purification and their cell number expansion. In the 2nd and 3rd year research project, investigators will optimize the 3-D cell culture model so as to increase the performances of CTC isolation/purification and proliferation. In the optimization process, investigators will explore the effect of cell culture model (e.g. static or perfusion cell culture, and 3-D cell culture using different 3-D scaffolding materials) or biochemical factors (e.g. glucose concentration, serum concentration, pH, or the supplements of growth factors/cytokines) on the the performances of CTC isolation/purification and proliferation.

SUMMARY:
The goal of this observational study is to validate and evaluate the clinical feasibility of using a 3-D cell culture model for CTCs isolation/purification and their cell number expansion in cancer patient with transitional cell carcinoma and patient without cancer.

This project first aims to study the clinical feasibility of utilizing a 3-D cell culture model for the isolation/purification of all possible CTCs in a blood sample in a label-free, viable, and high-purity manner. Through 3-D CTC culture, moreover, the cell number of CTCs can be adequately expanded. All these advantageous features are beyond what is currently possible by using the existing methods. In addition, the harvest of CTCs with above features is found valuable for the subsequent academic researches or clinical studies (e.g. molecular mechanisms underlying cancer metastasis, cancer-related gene mutation, biomarker discovery, and particularly CTCs-based chemotherapy drug testing). These could both facilitate and accelerate scientists to develop new therapeutic solutions for future cancer care.

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs), the rare cell species present in the blood, are considered to mainly contribute to cancer metastasis or relapse. Thus, the detection of CTCs is regarded as an essential clinical tool to detect metastatic cancer. Moreover, CTCs can be the therapeutic target of metastatic cancer care. Therefore, the use of viable CTCs as a biopsy to select therapeutic regimens (e.g. CTCs-based anti-cancer drug testing) opens up a promising route to realize personalized cancer therapy. With the recent advances in cell isolation or detection techniques, various novel approaches have been actively proposed to isolate/detect CTCs. Nevertheless, most of current methods might not be able to obtain the all possible, viable, and label-free CTCs with adequate cell purity and cell number for the subsequent CTCs-based anti-cancer drug testing or other bioassays. To tackle the above technical hurdles, the research project proposes the use of a specific 3-D cell culture technique for the isolation/purification, and cell number expansion of CTCs.

The working principle is based on our preliminary findings showing that the human leukocytes will die away in 3-D cell culture condition, whereas the CTCs will tend to aggregate and proliferate in such environment. Based on this phenomenon, the 3-D CTC cell culture can be used to isolate and purify the viable CTCs from the leukocyte background in a negative selection, and label-free manner, enabling the harvest of the all possible CTCs in a blood sample. Furthermore, the proliferation of CTCs in such 3-D cell culture can adequately expand the cell number of CTCs for the subsequent applications, which is currently impossible using the existing methods.

In the 1st year research project, investigators will further validate and evaluate the clinical feasibility of using a 3-D cell culture model for CTCs isolation/purification and their cell number expansion. In the 2nd and 3rd year research project, investigators will optimize the 3-D cell culture model so as to increase the performances of CTC isolation/purification and proliferation. In the optimization process, investigators will explore the effect of cell culture model (e.g. static or perfusion cell culture, and 3-D cell culture using different 3-D scaffolding materials) or biochemical factors (e.g. glucose concentration, serum concentration, pH, or the supplements of growth factors/cytokines) on the the performances of CTC solation/purification and proliferation. As a whole, investigators hope the proposed research project can find out an efficient and effective approach to isolate/purify/expand clinical CTCs in a viable, label-free, and high-purity manner. These harvested CTCs are valuable for the subsequent analytical tasks.

ELIGIBILITY:
Inclusion Criteria:

1. patients who agreed with the content of informed consent of the study protocol
2. patients who agreed the researcher to review the medical record
3. adults >20 years old
4. Patients have the right to asked withdrawing from the trial at any timepoints
5. meet the following requirements (1)cancer participants:cancer patients with transitional cell carcinoma (2)healthy participants:participants without cancer

Exclusion Criteria:

1. Patients who refused the collection of blood and the reviewing of medical record
2. The investigators suggest to withdraw

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cancer patients with transitional cell carcinoma
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
the effect of cell culture model for the Cell viability | baseline
  optimize the 3-D cell culture model to measure the Cell viability
the effect of cell culture model for the Cell viability | 3 month
  optimize the 3-D cell culture model to measure the Cell viability
the effect of cell culture model for the Cell viability | 6 month
  optimize the 3-D cell culture model to measure the Cell viability
the effect of cell culture model for the Cell number | baseline
  optimize the 3-D cell culture model to measure the Cell number
the effect of cell culture model for the Cell number | 3 month
  optimize the 3-D cell culture model to measure the Cell number
the effect of cell culture model for the Cell number | 6 month
  optimize the 3-D cell culture model to measure the Cell number

SECONDARY OUTCOMES:
the effect of biochemical factors for glucose concentration | baseline, pre-intervention
  investigate the effect of of biochemical factors to measure glucose concentration
the effect of biochemical factors for glucose concentration | 3 month
  investigate the effect of of biochemical factors to measure glucose concentration
the effect of biochemical factors for glucose concentration | 6 month
  investigate the effect of of biochemical factors to measure glucose concentration
the effect of biochemical factors for the serum concentration of growth factors/cytokines | baseline, pre-intervention
  investigate the effect of of biochemical factors to measure the serum concentration of growth factors/cytokines
the effect of biochemical factors for the serum concentration of growth factors/cytokines | 3 month
  investigate the effect of of biochemical factors to measure the serum concentration of growth factors/cytokines
the effect of biochemical factors for the serum concentration of growth factors/cytokines | 6 month
  investigate the effect of of biochemical factors to measure the serum concentration of growth factors/cytokines
the effect of biochemical factors for the serum pH | baseline
  investigate the effect of of biochemical factors to measure the serum pH
the effect of biochemical factors for the serum pH | 3 month
  investigate the effect of of biochemical factors to measure the serum pH
the effect of biochemical factors for the serum pH | 6 month
  investigate the effect of of biochemical factors to measure the serum pH

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Chih Kuo, Study Director — Ye,Siou-Ru
Locations (1):
- Chang Gung Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oppenheimer SB. Cellular basis of cancer metastasis: A review of fundamentals and new advances. Acta Histochem. 2006;108(5):327-34. doi: 10.1016/j.acthis.2006.03.008. Epub 2006 May 26. PMID 16730054
- [Background] Mehlen P, Puisieux A. Metastasis: a question of life or death. Nat Rev Cancer. 2006 Jun;6(6):449-58. doi: 10.1038/nrc1886. PMID 16723991
- [Background] Konstantopoulos K, Thomas SN. Cancer cells in transit: the vascular interactions of tumor cells. Annu Rev Biomed Eng. 2009;11:177-202. doi: 10.1146/annurev-bioeng-061008-124949. PMID 19413512
- See also: Cancer is a generic term for a large group of diseases that can affect any part of the body. Other terms used are malignant tumours and neoplasms. — http://www.who.int/mediacentre/factsheets/fs297/en/
- See also: This is the announcements about cancer in the website of Taiwan's DOH — http://www.hpa.gov.tw/BHPNet/Web/Index/Index.aspx